CLINICAL TRIAL: NCT03251235
Title: Neural Effects of Cognitive-behaviour Therapy in Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 09/H0604/55
Record Dates: First submitted 2017-07-31; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Panic Disorder
Keywords: cognitive behaviour therapy
MeSH Terms: conditions — Panic Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The care provider is not aware of whether a patient is allocated to the treatment group or the waiting group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Group receives four weekly sessions of CBT prior to experimental testing/ fMRI
  Interventions: Behavioral: Cognitive Behaviour Therapy
- Waiting Group (No Intervention): Group receives four weekly sessions of CBT after experimental testing/ fMRI

INTERVENTIONS:
Behavioral: Cognitive Behaviour Therapy
  Other Names: CBT
  Arms: Treatment Group

SUMMARY:
Exposure-based cognitive-behaviour therapy (CBT) for anxiety disorders is an effective intervention, but the brain mechanisms driving recovery are largely unknown. In this experimental medicine study, it will be investigated to what degree CBT affects neural markers of anxiety at an early stage of treatment, to identify dynamic mechanistic changes which might be crucial in the process of recovery as opposed to those seen following full treatment completion. Patients with panic disorder will be recruited and randomly allocated to a group receiving 4 weekly sessions of cognitive-behaviour therapy versus a waiting group not receiving any interventions until after the experimental procedure.

DETAILED DESCRIPTION:
PURPOSE The primary purpose is to enhance our understanding of the mechanisms essential in effective treatment of panic disorder.

METHODS Design: The present study has a between-subjects design, including a waiting group of participants with panic symptoms and a treatment group of participants with panic symptoms who will receive cognitive-behavioural treatment before being tested.

Participants: Twenty-eight volunteers with panic symptoms will be recruited. For participants who do meet the basic study criteria a phone screening appointment (10 - 30 mins) will be arranged to further screen for relevant inclusion and exclusion criteria. They will then be invited to the Department of Psychiatry for the pre-assessment session.

Treatment: Within the study, the investigators will offer participants a brief CBT course of 4 sessions, offered by the Lupina service. The Lupina Service forms part of the OBMH primary care Counselling & Psychology Service, based at the Warneford Hospital. It provides intensive individual CBT for panic disorder and agoraphobia and is staffed by trained graduate volunteer therapists. Potential therapists are psychology graduates with prior mental health experience, who are given 2 days' intensive training in CBT for panic disorder and agoraphobia by Alison Croft, Consultant Clinical Psychologist. They then receive group supervision of their clinical cases. Service evaluation indicates equivalent clinical outcomes for volunteer therapists relative to qualified clinical psychologists.

Procedure: Participants will be randomly allocated to either the treatment group or the waiting group. On arrival to the pre-assessment session, participants will be given a copy of the information sheet (previously seen during the online screening and e-mailed/ posted to them). They will be invited to fill out the consent form. Screening for past or previous psychiatric illness will be achieved using a structured clinical interview (SCID). In addition, participants will be asked to complete a battery of questionnaires. They will also be familiarised with the procedure occurring on the scanning day. Any outstanding questions the participant has will be addressed. The visit lasts about 1 to 1 ½ hrs. After the pre-assessment, a 4 weeks follow-up appointment (post-assessment) will be arranged with all participants. Half of the participants will be referred for treatment in the LUPINA group during that time. At the post-assessment 4 weeks later, the participants will be asked to come to the OCMR (Oxford Clinical Resonance Imaging) Department at the John Radcliffe Hospital. The visit will last a total of 2½ to 3 hrs and include a scanning session lasting 1 to 1 ½ hrs. Subjective mood will be assessed on the day of the scan using the State form of the State-Trait Anxiety Inventory, a Mood Visual Analogue Scale and the Positive and Negative Affect Schedule. In addition, subjects will again complete the questionnaires from the pre-assessment. After the scan, participants will work on two behavioural computer tasks using emotional faces and word stimuli to assess facial recognition and attention outside the scanner. At the end of the session, patients from the waiting group will be offered the taster-CBT treatment within the LUPINA service.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70
* Sufficiently fluent in English to understand the task and instructions
* PDSS score of at least 6
* At least two full panic attacks or limited symptoms attacks last 4 weeks

Exclusion Criteria:

* CNS-acting medication (antidepressants within last 6 months, benzodiazepine last 3 days)
* Current or past history of alcohol/ drug abuse
* Serious medical conditions (e.g., epilepsy, heart or respiratory problems)
* Done the task before
* Waiting group: under current psychotherapeutic treatment
* Pregnancy
* Contraindications to MRI e.g. pacemaker, mechanical heart valve, hip replacement, metal implants
* Severe claustrophobia that limits ability to participate in fMRI scanning

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-09-04 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Emotional processing | Treatment Group: post 4-week CBT treatment, waiting Group: post 4-week waiting
  Activation levels in the fear circuit of the brain in response to emotional stimuli (fMRI)

SECONDARY OUTCOMES:
Clinical symptom severity - Global anxiety and depression (self-report) | Baseline, after 4 weeks treatment/ waiting
  Hamilton Anxiety and Depression Scale HADS
Clinical symptom severity - Fear of physical sensations (self-report) | Baseline, after 4 weeks treatment/ waiting
  Body Sensations Questionnaire BSQ
Clinical symptom severity - Agoraphobic fear (self-report) | Baseline, after 4 weeks treatment/ waiting
  Agoraphobic Cognitions Questionnaire ACQ
Clinical symptom severity - Clinical severity and improvement (clinician-report) | Baseline, after 4 weeks treatment/ waiting
  Clinical Global Impression Scale CGI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Reinecke A, Thilo KV, Croft A, Harmer CJ. Early effects of exposure-based cognitive behaviour therapy on the neural correlates of anxiety. Transl Psychiatry. 2018 Oct 19;8(1):225. doi: 10.1038/s41398-018-0277-5. PMID 30341276